CLINICAL TRIAL: NCT06974942
Title: Investigation of Physical Activity in Adolescents Diagnosed With Familial Mediterranean Fever
Brief Title: Physical Activity in Adolescents With Familial Mediterranean Fever
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, PhD, Istanbul University - Cerrahpasa
Other Study IDs: paqfmf
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Familial Mediterranean Fever (FMF )
Keywords: Familial Mediterranean Fever; Physical Activity
MeSH Terms: conditions — Familial Mediterranean Fever; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Familial Mediterranean Fever: The study will include 76 patients diagnosed with Familial Mediterranean Fever who are being followed at the Division of Pediatric Rheumatology, Department of Pediatrics, Istanbul Faculty of Medicine, Istanbul University.
- Healthy control: The study will include healthy peers of adolescents diagnosed with FMF.

SUMMARY:
Familial Mediterranean Fever (FMF) is one of the most common autoinflammatory rheumatic diseases in childhood. Problems such as joint pain, muscle weakness, decreased aerobic capacity, and fatigue seen in children and adolescents with rheumatic disease may lead to low physical fitness levels. Limitation of physical performance is one of the possible consequences of chronic diseases that occur during childhood. At the same time, children with chronic illness face many challenges in participating in physical activity. Pediatric patients with rheumatic diseases tend to be physically inactive and, compared to their healthy peers, generally avoid participating in physical activity due to the limitations imposed by the disease. Often, the disease itself paves the way for decreased functional capacity and the development of deconditioning. Therefore, prescribing physical activity and exercise to pediatric populations with chronic illnesses is of great importance. This approach helps alleviate both the symptoms related to chronic diseases and the lifelong complications secondary to pharmacological treatments, and also prevents the development of new chronic conditions.

Participation in adequate physical activity is one of the most important behaviors individuals can adopt to maintain their health and well-being. Globally, public health physical activity guidelines address the exercise needs of children and adolescents. The European Alliance of Associations for Rheumatology (EULAR) highlights in its physical activity and exercise guidelines for patients with rheumatic diseases that the physical activity recommendations made for the general population are also applicable to patients with rheumatic diseases.

With this cohort study, it is aimed to examine physical activity (PA) in detail in adolescents diagnosed with FMF and to compare them with healthy peers. This study is one of the first in our country to provide comprehensive data on the PA levels of adolescents with FMF. The findings obtained will contribute to understanding PA levels and exercise perception, and guide the planning of exercise programs to be developed for these individuals. Moreover, the results of the study may also serve as a basis for future research in children and adolescents with various chronic diseases, especially those with FMF.

ELIGIBILITY:
Inclusion criteria for patients with FMF:

* Be between 12-18 years of age
* Have been diagnosed with FMF for at least 6 months at the Pediatric Rheumatology Department of Istanbul Faculty of Medicine
* Be undergoing routine medical treatment for FMF
* Be willing to participate in the study

Exclusion criteria for patients with FMF:

* Adolescents whose participation in the study is not wanted by their family
* Having vestibular or neurological balance problems
* Presence of scoliosis, leg length discrepancy, or recent lower extremity surgery
* Adolescents with visual or hearing impairments

Inclusion criteria for healthy peers:

* Be between 12-18 years of age
* Be willing to participate in the study

Exclusion criteria for healthy peers:

* Adolescents whose participation in the study is not wanted by their family
* Having vestibular or neurological balance problems
* Presence of scoliosis, leg length discrepancy, or recent lower extremity surgery
* Adolescents with visual or hearing impairments

Exclusion criteria for removal:

- Leaving at least 3 questions unanswered in the questionnaires

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Our study consists of two cohorts, where the physical activity level, physical activity competence, and motivation for physical activity of adolescents with Familial Mediterranean Fever (FMF) will be evaluated and compared with their healthy peers.
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Adolescent Physical Activity Questionnaire (PAQ-A) | Baseline
  The Adolescent Physical Activity Questionnaire, developed by Kowalski and colleagues in 1997 to assess the physical activity levels of high school students, is an 8-item, 5-point Likert scale tool based on recalling the past 7 days. The 8 items in the scale are used to calculate the physical activity score. The 9th item inquires whether the participant was ill during the past week or if there was any condition preventing normal physical activity. However, this item is not included in the scoring.
  The first item lists 24 types of physical activity. The frequency of each activity is scored as "never" (1 point), "1-2" (2 points), "3-4" (3 points), "5-6" (4 points), or "7 or more times" (5 points). The result is divided by 24 to obtain the activity score for this item. For items 2-7, responses start with the lowest level of physical activity (1 point) and increase to the highest level (5 points). Item 8 evaluates the frequency of physical activity over the 7 days of the week. Responses a

SECONDARY OUTCOMES:
Physical Activity Participation Motivation Scale | Baseline
  This scale was developed to assess the motivation of high school students to participate in physical activity. It is a 16-item scale consisting of three factors: individual reasons, environmental reasons, and lack of reasons. In the study, the scale items are rated using a 5-point Likert scale: "Strongly disagree," "Disagree," "Undecided," "Agree," and "Strongly agree." The lowest possible score on the scale is 16, and the highest score is 80. Higher scores indicate more positive motivation to participate in physical activity.
  In this context, the scores on the Physical Activity Participation Motivation Scale are interpreted as follows: 1-16 indicates very low motivation, 17-32 indicates low motivation, 33-48 indicates medium motivation, 49-64 indicates high motivation, and 65-80 indicates very high motivation for physical activity participation. Items 3, 9, 13, 14, 15, and 16 are reverse-scored. The Cronbach alpha values range from 0.82 to 0.89, indicating good reliability.
Physical Activity Competence Scale | Baseline
  Physical Activity Competence Scale (PACS), adolescents' physical activity competence in different physical activity areas (at school, in transportation, at home, leisure and recreation, and school-based walking and transportation) is a 5-dimensional and 26-item scale developed to assess their competence.
  PACS consists of 5 dimensions and 26 items (At school: 6 items, In transportation: 3 items, At home: 5 items, Leisure and recreation: 6 items, School-based walking and transportation: 6 items). The scale form consists of two parts. The first part contains demographic information, and in the second part, participants are asked how confident they are in participating in physical activities in the five physical activity areas. A 10-point Likert-type scale (0 = "I have no confidence" and 100 = "I have full confidence") is used for the items. The total average score is calculated from the answers to the items in each domain and ranges between 0 and 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No